CLINICAL TRIAL: NCT04038983
Title: Risk for Short-term Adverse Events in Older Users in the Emergency Department: An Observational Cohort Study on Evaluation of PRISMA-7
Brief Title: Risk for Short-term Adverse Events in Older Users in the Emergency Department
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1852
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Old Age; Medical Care; Survey
Keywords: Emergency, Old patients , Survey Questionnaire
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: ER2 is a simple and standardized clinical tool composed of two sequential components: an assessment followed by recommendations for intervention. The assessment component of ER2 consists of 6 very simple closed-ended format questions (i.e., yes versus no) which are: Age category (≥ 85), male, polypharmacy (≥ 5 different medications per day), use of formal (health care or social professional) and/or informal (family and/or friend) home support, use of a walking aid regardless of its type, and temporal disorientation (inability to give the current month and/or year). A score of five points is assigned to the items "use of walking aid" and "temporal disorientation", whereas, for the other items, the assigned score is one point. The weighting of points for ER2 items is based on the results of our previous studies (21-24). Scores range from 0 (lowest risk) to 14 (highest risk). ER2 scores stratify the risk for short-term ED adverse events into three levels: low, moderate and high.

SUMMARY:
The study evaluates the performance criteria of abnormal PRISMA-7 score, length of stay in Emergency department and in hospital, and hospital admission in older Emergency department users.

DETAILED DESCRIPTION:
In Quebec, Canada, the "Program of Research on Integration of services for the Maintenance of Autonomy" (PRISMA-7) is the Ministry of Health and Social Services' reference tool for the frailty assessment of older Emergency department users. This tool has been initially developed and validated to assess disabilities in older community dwellers with the aim to quickly identify older individuals at risk for disabilities and who should undergo a comprehensive assessment. PRISMA-7 has a high sensitivity for identifying frailty in older community dwellers but its performance criteria for this goal has never been examined in older Emergency Department users. Recently, a systematic review underscored that PRISMA-7 has all characteristics for being a usable clinical tool in Emergency department because it is a brief (i.e., <5 min), simple and multidimensionality assessment. PRISMA-7 is composed of 7 questions assessing health and functionality of older adults and stratifies risk for disability in two levels: low versus high. PRISMA-7 is a prognostic tool for disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the ER2 study( Emergency Room Evaluation and Recommendation)
* Having a score test of Prisma 7( Program of Research on Integration of Services for the Maintenances of Autonomy) at Emergency.

Exclusion Criteria:

* Never being enrolled in the ER2 study( Emergency Room Evaluation and Recommendation)
* Never having a score test of Prisma 7( Program of Research on Integration of Services for the Maintenance of Autonomy) at Emergency

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: There are two survey questionnaires that will be fill out by nurses when a patient who are 75 years old and over arrives: Prisma-7 ( Program of Research on Integration of Services for the Maintenances of Autonomy) and ER2 ( Emergency Room Evaluation and Recommendation).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | around 12 months
  The length of hospital stay is defined as the average number of days that patients spend in hospital. It will be used the ER2 tool ( Emergency Room Evaluation and Recommendation) to calculate the length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada